CLINICAL TRIAL: NCT00291421
Title: International Outcomes Survey In Dementia (IOSID)
Brief Title: A Survey Study of the Treatment and Outcome Management in Patients Diagnosed With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Other Study IDs: CR003937
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Alzheimer Disease; Dementia; Nervous System Diseases; Mental Disorders; Brain Diseases
Keywords: Alzheimer's Disease; Dementia; Brain Disease; Memory Loss; Caregiver; Primary Caregiver; Observation; galantamine; donepezil; rivastigmine; Quality of life
MeSH Terms: conditions — Alzheimer Disease; Dementia; Nervous System Diseases; Mental Disorders; Brain Diseases; Memory Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to collect and compare information regarding the treatment and outcome of patients diagnosed with Alzheimer's disease who are receiving either drug or nondrug treatment. Information will be collected from patients and their primary caregivers.

DETAILED DESCRIPTION:
Dementia is a chronic, progressive brain disease that may involve a number of symptoms, including memory loss and changes in personality, behavior, judgment, attention span, language and thought. The most common type of dementia is Alzheimer's disease. Over time, patients with Alzheimer's disease may lose ability to perform daily tasks related to personal care (for example bathing, dressing, eating) and may be unable to handle money or travel to familiar places. Dementia is one of the main reasons people are admitted to long-term care in residential or nursing homes.Treatments or services that prevent or delay admission into these institutions are important because they may help decrease or delay the use of health or social care resources that are increasing in a growing elderly population.This study is a large-scale survey that will provide information related to the treatment of Alzheimer's disease, including information regarding treatment patterns, characteristics of patients with Alzheimer's disease, estimates of costs of care, disease outcomes, patients' ability to function daily and quality of life for caregivers. This study will examine the current management of patients with mild and moderate Alzheimer's disease in real life settings. As opposed to a clinical trial in which a particular group of patients is selected to participate and where treatments may be specified and possibly compared with a placebo (an inactive substance), this study will include a wider variety of patients and treatment options to more closely represent the management of Alzheimer's disease in current clinical practice. Information will be collected from patients in Europe and other countries who are being treated by a doctor for mild to moderate Alzheimer's disease. Patients receiving treatment with one of the following medications approved for treatment of Alzheimer's disease (galantamine, donepezil, rivastigmine or tacrine) and patients receiving nondrug treatment (disease progression monitoring, ginkgo extracts, Vitamin E, estrogen, etc) may participate. No treatment or procedures will be specified and no medication will be provided by the Sponsor of this study. Treatment of Alzheimer's disease may be stopped, started or changed by the patients' individual doctors as appropriate. Information regarding disease status, treatment, behavior, ability to function and use of social care services (day care, home care, meals on wheels, social work) will be collected from patients. Information regarding quality of sleep of the patient and caregiver, amount of care required by the patient and well-being/general quality of life will be collected from caregivers. Information will be collected every 6 months for a period of 2 years, with a possible additional follow-up period of 2 years. If a patient in the study dies, the collection of information will stop. If a patient in the study is permanently admitted to a supported care, nursing home or residential care facility, collection of information will stop but follow-up with the caregiver will be conducted at the end of the 2-year survey to determine if the patient is alive or deceased. The study hypothesis is that treatment of Alzheimer's disease with medication may improve patient status, reduce caregiver dependency, improve caregiver quality of life, reduce the amount of social care services needed and prolong or prevent admission to long-term institutions of patients with Alzheimer's disease Since the study involves only collection of information, no treatment will be required by the Sponsor and no medication will be supplied by the Sponsor

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with new or previous mild or moderate Alzheimer's disease diagnosed by a doctor according to medically-accepted definitions
* Patients living in ordinary households (for example in their own home or in the home of a family member or friend, not in nursing homes or other long-term care facilities)

Exclusion Criteria:

* Patients who are currently participating in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2360 (Actual)
Dates: Start 2002-07; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.